CLINICAL TRIAL: NCT05955248
Title: A Novel Multimodal Intervention for Surgical Prehabilitation of Patients With Lung Cancer: the MMP-LUNG Trial
Brief Title: Multimodal Prehabilitation for Lung Cancer Surgery
Acronym: MMP-LUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stéphanie Chevalier (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Stéphanie Chevalier, Associate Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MUHC REB 2022-7782
Record Dates: First submitted 2023-06-22; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer; Surgery
Keywords: Prehabilitation; Nutritional Supplement
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, 3 parallel arms (multimodal intervention, MM; nutritional supplement, NUT; control, CTRL), double-blind and placebo-controlled for supplement, single centre.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinding of exercise is not possible therefore participants will be aware if they are in the MM group. However, research personnel performing outcome assessments will be blinded to group allocation. Groups CTRL and NUT will be double-blinded. Supplements will be packaged by the supplier in coded-labeled sachets (for powder) and bottles (for oil). The supplier will disclose the code to a research person not associated with the trial. Research staff will prepare boxes of supplements (or placebo) according to coded group allocation. All participants will be instructed to not self-supplement with commercially available products, to minimize the risk of group contamination. All data and biological samples will be coded such that participant's identification will not be disclosed to research personnel conducting analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (CTRL) (Placebo Comparator): Participants will be treated following Enhanced Recovery After Surgery (ERAS) protocols + placebo supplements containing maltodextrin and sunflower oil
  Interventions: Dietary Supplement: Placebo Control (CTRL)
- Mixed-nutriend supplement (NUT) (Active Comparator): Mixed nutrient supplement containing whey protein, leucine, vitamin D and omega 3 fatty acids
  Interventions: Dietary Supplement: Mixed-nutriend supplement (NUT)
- Multi-modal intervention (MM) (Active Comparator): Multimodal prehabilitation including structured exercise (1 supervised exercise session per week + home-based exercise program), nutritional optimization with dietician, NUT intervention, and relaxation strategies.
  Interventions: Dietary Supplement: Mixed-nutriend supplement (NUT); Other: Multimodal Prehabilitation (MM)

INTERVENTIONS:
Dietary Supplement: Mixed-nutriend supplement (NUT) — Participants will follow ERAS protocol and will receive dietary counselling and anxiety management counselling as needed. They will receive the active multi-nutrient supplement made of whey protein + leucine + vitamin D doses pre-mixed in unlabeled packets prepared by Gruppo Nutrition to dilute in a cup (250 mL) of water. In addition, participants will ingest 15 mL of fruit-flavored fish oil, provided as a liquid oil. They will receive a dosing cup, pre-marked to 15 mL, for a total dose providing 2120 mg eicosapentaenoic acid (EPA) and 1320 mg docosahexaenoic acid (DHA).
  Arms: Mixed-nutriend supplement (NUT); Multi-modal intervention (MM)
Other: Multimodal Prehabilitation (MM) — Participants will follow ERAS protocol and will receive dietary counselling and anxiety management counselling as needed. They will receive the NUT intervention + structured exercise training prescribed by a kinesiologist (1. 30 min of aerobic exercise per day of their preferred type (ex. walking) and 2. 30 min of resistance exercise targeting major muscle groups, every second day for 2 sets of 8-12 reps). Training will be performed for 4 weeks prior to surgery (1x/week supervised by kinesiologist at hospital, 2x/week at alone at home)
  Arms: Multi-modal intervention (MM)
Dietary Supplement: Placebo Control (CTRL) — Participants will follow ERAS protocol and will receive dietary counselling and anxiety management counselling as needed. They will receive a placebo dietary supplement made of maltodextrin and sunflower oil.
  Arms: Control (CTRL)

SUMMARY:
The main objective of this randomized controlled trial (RCT) is to investigate whether a multimodal prehabilitation intervention combining a mixed-nutrient supplement with structured exercise training (MM) or the supplement alone (NUT), against a placebo (CTRL), leads to improvement in functional capacity and postoperative outcomes in surgical patients with lung cancer, at nutritional risk. This will be tested in a single centre RCT of 3 parallel arms, double-blinded for the supplement. Female and male participants (n=168, >=45 y) will be randomized to a 10-week intervention spanning 4 weeks pre-surgery and 6 weeks post-hospital discharge. The primary outcome is functional capacity as measured by the 6-minute walk test. Secondary outcomes include muscle mass, quality and strength, quality of life, length of hospital stay, and postoperative complications.

DETAILED DESCRIPTION:
RATIONALE: The preoperative period is an opportune time to actively engage and empower patients in improving their functional, nutritional and mental status in anticipation of the surgical stress. Considering that lung cancer patients often present with poor nutritional status and physical function prior to surgery, providing a nutritional supplement to increase protein, leucine, vitamin D and omega-3 fatty acid FA intake with a structured exercise program and relaxation techniques should improve muscle mass, strength and physical performance.

MAIN OBJECTIVE: to test the effect of a multimodal RCT prehabilitation intervention (MM) combining a mixed-nutrient supplement with structured exercise training or the supplement alone (NUT) against a placebo (CTRL), on functional pre- and postoperative outcomes in surgical patients with lung cancer at nutritional risk.

STUDY DESIGN: 10-week randomized controlled trial of 3 parallel arms, double-blinded for supplement: control (CTRL), multi-nutrient supplement (NUT) and multimodal intervention (MM). After baseline assessment, patients will be randomized to either group in a 1:1:1 CTRL:NUT:MM ratio using a computer-generated randomization scheme by permuted block sizes, with stratification by sex and functional capacity (< or > 450 m on the 6-minute walk test (6MWT). Consecutive adult patients = or > 45 years scheduled for elective video-assisted thoracic surgery or open thoracotomy surgery of non-small cell lung cancer (NSCLC) stages I, II or IIIa and a Patient-Generated Subjective Global Assessment (PG-SGA) score = or > 3, will be approached following their first appointment with their surgeon at the McGill University Health Centre (MUHC)-Montreal General Hospital.

INTERVENTION: The NUT arm will ingest a multi-nutrient supplement consisting of whey protein + leucine + viatmin D, and fish oil. The CTRL participants will receive placebo supplements with the same physical aspect, flavor and packaging as the active supplement.The MM arm will receive the NUT intervention in addition to performing structured exercise and relaxation techniques for 4 weeks prior to surgery and 6 weeks after hospital discharge.

OUTCOMES: Primary: physical capacity measured by the 6MWT; Secondary: physical function, muscle strength, total skeletal muscle mass, leg muscle volume and density, body composition, quality of life, length of stay and post-operative complications; Other: dietary intake, physical activity, exercise tolerance, pulmonary function, clinical markers.

STATISTICAL ANALYSIS: Intention-to-treat analysis will be performed in the primary analyses. For preoperative data, analysis of covariance (ANCOVA) will compare between-group differences at 4-week preoperative time, conditioned for baseline data, including predefined covariates in the model (age, sex, BMI). The hypothesis of full recovery from the intervention at 6 weeks postoperative (i.e. 6MWT returning back to or exceeding baseline) will be tested by logistic regression (yes/no). Between-group changes in other outcomes will be evaluated as differences in mean or proportions, as appropriate, with 95% CIs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45 years and over
* Diagnosed with NSCLC stages I, II or IIIa and scheduled for video-assisted thoracic surgery (VATS) or open thoracotomy surgery for cancer resection
* At nutritional risk (defined as Patient Generated-Subjective Global Assessment score = or >3)

Exclusion Criteria:

* Prior recent (<2 months) adjuvant therapy (chemo- or radio-therapy)
* Inability to perform, or comorbidities contraindicating, exercise (defined as CPET <10 mL O2/kg/min)
* Unable to walk (uses a wheelchair)
* Allergy to milk or seafood
* Hypercalcemia (total serum Ca >2.60 mmol/L or ionized Ca >1.30 mmol/L)
* Hypervitaminosis D (serum 25(OH)D >375 nmol/L)
* Glomerular filtration rate (<30 mL/min/1.73m2)
* Insufficient understanding of English or French to provide informed consent

Patients taking omega-3 FA supplements will be asked to withhold them during the study; those taking vitamin D will continue unless baseline serum 25(OH)D >80 nmol/L.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in preoperative functional walking capacity | From baseline (4 weeks pre-surgery) to surgery
  6-Minute walking test (6MWT): measured as the distance walked during 6 minutes, along a 20-m corridor, expressed in meters
Postoperative functional walking capacity | 6 weeks after surgery
  6-Minute walking test (6MWT): measured as the distance walked during 6 minutes, along a 20-m corridor, expressed in meters

SECONDARY OUTCOMES:
Change in handgrip strength | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Handgrip strength using hand-held Jamar dynamometer, measured in kg
Change in total skeletal muscle mass | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Estimated using deuterium-labeled creatine (D3-creatine), measured in kg
Change in foreleg muscle surface area | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Skeletal muscle surface area will be measured in the dominant foreleg, using peripheral quantitative computerized tomography (pQCT, Stratec XCT2000), measured in cm2.
Change in foreleg myosteatosis (radiodensity) | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Skeletal muscle radiodensity will be measured in the dominant foreleg, using peripheral quantitative computerized tomography (pQCT, Stratec XCT2000), measured in mg/cm3.
Change in body weight and composition | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Soft lean and fat mass measured by bioelectrical impedance (seca mBCA 515)
Change in self-reported quality of life | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Measured by the 36-item Short Form Survey (SF36, score 0-100; higher means better quality of life)
Change in self-reported functional assessment | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Measured by the Functional Assessment of Cancer Therapy - Lung questionnaire (FACT-L score 0-136, higher means better quality of life)
Length of hospital stay | 6 weeks after surgery
  Recorded from medical charts, expressed in days
Number and severity of postoperative complications | 6 weeks after surgery
  Recorded from medical charts and graded by severity following the Clavien-Dindo classification

OTHER OUTCOMES:
Change in dietary intake | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Collected from 3-day food diaries, using a mobile application (Keenoa)
Change in plasma phospholipid fatty acid profile | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Plasma lipids will be extracted with organic solvents, phospholipids isolated on thin-layer chromatography, and FAs methylated for determination by gas chromatography-flame-ionization analysis. Change in long-chain omega-3 fatty acids will be used as an objective measure of adherence to fish oil supplement.
Change in serum vitamin D 25(OH)D concentrations | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Concentrations will be measured by the MUHC-Central Lab. Used as an objective measure of adherence to the supplement.
Change in serum C-Reactive Protein (CRP) | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Measured as high-sensitive CRP by the MUHC-Central Lab.
Change in serum albumin | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Analyzed by standard procedures at the MUHC-Central Lab
Change in serum pre-albumin | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Analyzed by standard procedures at the MUHC-Central Lab
Change in serum hemoglobin | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Analyzed by standard procedures at the MUHC-Central Lab
Change in complete blood count | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Analyzed by standard procedures at the MUHC-Central Lab
Change in preoperative exercise tolerance | From baseline (4 weeks pre-surgery) to surgery
  Assessed as oxygen consumption during cardiopulmonary exercise testing (CPET) at anaerobic threshold and peak exercise, in mL O2/kg/min
Change in forced expiratory volume (FEV1) | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Spirometry standard methods to measure the forced expiratory volume (FEV1)
Change in forced vital capacity (FVC) | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Spirometry standard methods to measure the forced vital capacity (FVC) and calculate FEV1/FVC ratio.
Change in self-reported physical activity level score | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Measured with the Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire, score 0 - x (no maximum score), higher mean more activity.
Change in physical activity | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Measured by accelerometry (Actigraph wGT3X-BT) during the intervention. Step count and time spent at sedentary, light, moderate/ vigorous activity, and sleeping time will be recorded.
Change in anxiety/depression score | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  Hospital Anxiety and Depression Scale (questionnaire). Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Change in Patient-Generated Subjective Global Assessment (PG-SGA) score | From baseline (4 weeks pre-surgery) to 6 weeks after surgery
  PG-SGA questionnaire, total score. A higher score indicates higher nutritional risk or malnutrition.
Number of adverse events | Through study completion, an average of 10 weeks
  Any adverse event, related or not to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Chevalier, PhD, Principal Investigator — McGill University
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Moyen A, Fleurent-Gregoire C, Gillis C, Zaks R, Carli F, Scheede-Bergdahl C, Spicer J, Cools-Lartigue J, Najmeh S, Morais JA, Mazurak V, Chevalier S. Novel multimodal intervention for surgical prehabilitation on functional recovery and muscle characteristics in patients with non-small cell lung cancer: study protocol for a randomised controlled trial (MMP-LUNG). BMJ Open Respir Res. 2025 May 22;12(1):e002884. doi: 10.1136/bmjresp-2024-002884. PMID 40404185